CLINICAL TRIAL: NCT01891370
Title: Median Study for Biochemical Serum Markers in First Trimester of Pregnancy
Status: Completed | Type: Observational
Sponsor: PerkinElmer, Wallac Oy (Industry)
Responsible Party: Sponsor
Other Study IDs: 11060
Record Dates: First submitted 2013-06-28; First posted 2013-07-03 (Estimated); Last update posted 2015-09-28 (Estimated); Status verified 2015-09

CONDITIONS: Pregnancy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Serum
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to get initial values (normal medians) for certain biochemical serum markers for pregnancy weeks 10-13. Also initial values for mean arterial blood pressure measurement and certain ultrasound measurement may be established.

ELIGIBILITY:
Inclusion Criteria:

* written informed consent
* maternal age 18 - 45 years
* gestational age 10 -13 (+6 days)verified by ultrasound

Exclusion Criteria:

* mental retardation or other mental disorders that impose doubts regarding the true subject's willingness to participate in the study
* lack of needed demographic data

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: women in first trimester of pregnancy coming to antenatal assessment
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2013-07; Primary Completion 2014-12 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
levels of biochemical serum markers | 10-13 wks gestation

CONTACTS AND LOCATIONS:
Locations (3):
- Hospital Tuanku Jaafar, Seremban, Malaysia
- MCU-FDT Medical Foundation, Caloocan, Philippines
- Khon Kaen University, Khon Kaen, Thailand